CLINICAL TRIAL: NCT04596878
Title: A Multi-centre Study to Evaluate the Safety, Tolerability and Immunogenicity of Two Doses of a Group B Streptococcus Vaccine (GBS-NN/NN2) in Women Who Are Pregnant and Living With HIV and Women Who Are Pregnant and do Not Have HIV
Brief Title: Study of a Group B Streptococcus Vaccine in Pregnant Women Living With HIV and in Pregnant Women Who do Not Have HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minervax ApS (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MVX0005
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Group B Streptococcal Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Intervention Model Description: Randomised, placebo controlled, double-blind, parallel group, multicentre study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GBS-NN/NN2 in pregnant women living with HIV (Experimental): 2 doses of 0.5mL intramuscular injection GBS-NN/NN2 containing 50 µg GBS-NN and 50 µg NN2 administered 28 days apart in pregnant women living with HIV
  Interventions: Biological: GBS-NN/NN2
- Placebo Comparator in pregnant women living with HIV (Placebo Comparator): 2 doses of 0.5mL intramuscular injection 0.9% normal saline administered 28 days apart in pregnant women living with HIV
  Interventions: Biological: Placebo
- GBS-NN/NN2 in pregnant women who do not have HIV (Experimental): 2 doses of 0.5mL intramuscular injection GBS-NN/NN2 containing 50 µg GBS-NN and 50 µg NN2 administered 28 days apart in pregnant women who do not have HIV
  Interventions: Biological: GBS-NN/NN2
- Placebo Comparator in pregnant women who do not have HIV (Placebo Comparator): 2 doses of 0.5mL intramuscular injection 0.9% normal saline administered 28 days apart in pregnant women who do not have HIV
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GBS-NN/NN2 — GBS-NN/NN2 bound to Alhydrogel as an adjuvant.
  Arms: GBS-NN/NN2 in pregnant women living with HIV; GBS-NN/NN2 in pregnant women who do not have HIV
Biological: Placebo — Normal Saline 0.9%
  Arms: Placebo Comparator in pregnant women living with HIV; Placebo Comparator in pregnant women who do not have HIV

SUMMARY:
A randomised, placebo-controlled, double-blind study to evaluate the safety, tolerability and immunogenicity of the GBS-NN/NN2 (Recombinant protein vaccine against Group B Streptococcus) vaccine in women living with HIV and women without HIV,and their newborn babies from vaccination up to delivery/birth. Mothers and babies will be followed up for 6 months post-delivery.

DETAILED DESCRIPTION:
100 women who are pregnant and living with HIV will randomly receive two 0.5 mL (millilitre) intramuscular injections of GBS-NN/NN2 vaccine (60 women) or placebo (15 women).

100 women who are pregnant and do not have HIV will randomly receive two 0.5 mL intramuscular injections of GBS-NN/NN2 vaccine (60 women) or placebo (15 women).

Participants will be screened at 24 to 28 weeks gestation (Days -14 to Day -1) and the groups will be dosed in parallel. The first dose of vaccine or placebo will be administered at Day 0 and the second dose will be administered 28±2 days later. Delivery is anticipated to be approximately 10 to 14 weeks after the first dose of vaccine.

For the analysis of the immune response, the placebo groups will be combined. For safety, the placebo groups will be analysed separately and will be combined for comparison with the potential vaccine groups.

ELIGIBILITY:
Inclusion Criteria:

1. Participants at least 18 years old and not older than 40 years of age.
2. Pregnant women who are between 26 weeks and 30 weeks (inclusive) gestation on the planned day of vaccination with a singleton, uncomplicated pregnancy. Gestational age to be determined on the following hierarchal basis with guidance to the GAIA (Global Alignment of Immunisation Safety Assessment in pregnancy) criteria:

   1. ultrasound estimate of gestational age,
   2. date of last menstrual period
   3. fundal height
3. HIV status to be based on rapid, confirmatory test, unless a documented test of the participant being sero-positive for HIV and history documented in the notes.
4. Women living with HIV, HIV viral load <1000, on antiretroviral therapy for at least 3 months prior to screening and clinically well.
5. Expected to be available for the scheduled clinic visits for the duration of the study, agree to be contacted by telephone during study participation, and is willing to give parental consent for her infant to participate in the study

Exclusion Criteria:

1. Women who are HBSAg and/or HCV (hepatitis C virus) positive
2. Women who test positive for syphilis as per standard testing
3. Women knowingly carrying, at screening, a malformed or genetically abnormal foetus based on ultrasound
4. Women who have experienced a previous stillbirth prior to going into labour
5. Women with placenta previa
6. Women with documented chronic or pregnancy induced hypertension at screening
7. Women with 1+ protein in urine and hypertension defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) at ≥20 weeks of gestation in a woman with a previously normal blood pressure
8. Women with >1+ of protein in urine (regardless of blood pressure)
9. Women with gestational, type 1 or type 2 diabetes.
10. Women with glycosuria on dipstick
11. Women known to be allergic to any components of the vaccine, who are known to be allergic to aluminium or have had an allergic reaction to any previous vaccination.
12. Women with HIV viral load >1000 at screening.
13. Women living with HIV who have been on antiretroviral therapy for less than 3 months prior to screening. (Women who are diagnosed with HIV between screening and dosing will not be eligible.)
14. Women with history or presence of significant cardiovascular disease, pulmonary, hepatic, gallbladder or biliary tract, renal, haematological, gastrointestinal, endocrine, immunologic, dermatological, neurological, psychiatric, autoimmune disease, cognitive disorder or current infection and significant illness 4 weeks prior to randomization.
15. Women with current or history of drug or alcohol abuse within the last two years.
16. Women who have received a vaccine within 28 days of receiving the first dose of GBS NN/NN2 or placebo or who expect to require vaccination during the course of the study. (Vaccines recommended for administration during pregnancy e.g. tetanus toxoid, pertussis and influenza are permitted. Administration of concurrent vaccines must not be within 7 days of investigational vaccine.)
17. Women who have a fever (axillary temperature >37.9°C) on the day of dosing or have had an acute infection in the 7 days before dosing.
18. Women who have any bleeding disorders that prolong the bleeding time.
19. Women who are receiving immunosuppressive medication, including systemic steroids (inhaled and topical steroids are acceptable).
20. Women who have received blood or blood products and/or plasma derivatives or any immunoglobulin preparations in 12 weeks preceding screening.
21. Women with severe anaemia, haemoglobin < 9g/dL (90 g/L) as per Sheffield grading system ( > Grade 1)
22. Women who are currently breast feeding
23. Women who are part of the study personnel or a close family member of study personnel.
24. Women who in the opinion of the investigator are not suitable to participate in the study.
25. Concurrent participation in another clinical trial during which subject will be exposed to an investigational product .

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 205 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | From vaccination up to delivery/birth
  Adverse events
Gestational age of newborn baby | At birth
  Gestational age of newborn baby
Weight of newborn baby | At birth
  Weight of newborn baby
Length of newborn baby | At birth
  Length of newborn baby
Head circumference of newborn baby | At birth
  Head circumference of newborn baby
Apgar score for newborn baby | At birth
  Apgar score for newborn baby
IgG (Immunoglobulin G) antibody concentration | At birth
  IgG antibody concentration specific to the GBS-NN/NN2 vaccine measured in maternal blood and cord blood

SECONDARY OUTCOMES:
Incidence of significant adverse reactions in mothers | From delivery to 6 months post-delivery
  Significant adverse reactions
Developmental milestones of babies | At 6 months
  Milestones assessed using ages and stages questionnaires
Geometric mean antibody concentration | At 4 weeks post first injection and at 4 weeks post second injection
  Geometric mean antibody concentration
Geometric mean antibody concentration of cord and maternal blood | At delivery
  Geometric mean antibody concentration of cord (or newborn blood within 48 hours of birth) and maternal blood
Geometric mean fold increase in antibody concentration in maternal blood | At 4 weeks post first injection and at 4 weeks post second injection
  Geometric mean fold increase in antibody concentration in maternal blood
Geometric mean fold increase in antibody concentration in maternal blood | From baseline to delivery
  Geometric mean fold increase in antibody concentration in maternal blood
Proportion of mothers and newborn babies achieving vaccine specific IgG antibody concentrations | At delivery
  Proportion of mothers and newborn babies achieving vaccine specific IgG antibody concentrations in maternal and cord blood samples respectively, above pre-defined arbitrary thresholds.

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Kitson, Study Director — gkitson@propharmapartners.uk.com
Locations (3):
- South Africa (2):
  - Empilweni Services and Research Unit (ESRU), Rahima Moosa Mother and Child Hospital, Johannesburg
  - University of the Witwatersrand, Johannesburg (Respiratory and Meningeal Pathogens Research unit), Johannesburg
- MUJHU Research Collaboration/MUJHU Care Ltd, Kawempe National Referral Hospital, Kawempe, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galiza EP, Khalil A, Heath PT. Update on Vaccines in Antenatal Care. Pediatr Infect Dis J. 2024 Feb 1;43(2):e60-e62. doi: 10.1097/INF.0000000000004183. Epub 2023 Dec 27. No abstract available. PMID 38190492